CLINICAL TRIAL: NCT06659874
Title: Investigation of the Relationship Between Core Muscles Functions and Symptoms of Patients with Abdominal Bloating/Distension
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Collaborators: Ege University Medical School (Other); The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Melahat AKTAŞ, Research assistant, Dokuz Eylul University
Other Study IDs: 2022/35-14
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-04

CONDITIONS: Bloating; Distension
Keywords: abdominal bloating/distension; core muscles; electromyography
MeSH Terms: conditions — Dilatation, Pathologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to investigate the relationship between core muscle functions (strength, endurance, thickness) and symptoms in individuals with abdominal bloating/distension. The main questions it aims to answer are:

Does symptoms in individuals with abdominal bloating/distension have an effect on core muscles? How do core muscles change based on an increase or decrease in these symptoms?

DETAILED DESCRIPTION:
In studies on individuals with abdominal bloating/distension in the literature, the diaphragm, abdominal muscles, and pelvic floor muscles have been examined separately. There is no study that examines all core muscles together in such cases. Additionally, there is no study examining the relationship between core muscle function and symptoms. Therefore, the aim of our study is to investigate the relationship between core muscle functions (strength, endurance, thickness) and symptoms in individuals with abdominal bloating/distension.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of abdominal bloating/distension made by a physician according to the Rome IV Criteria
* Be female between 18 and 65 years of age
* Volunteer to participate"

Exclusion Criteria:

* Having a serious neurological, pulmonary, systemic, orthopedic, or metabolic disease accompanying bloating-distension
* Being under 18 or over 65 years of age
* Being pregnant
* Having any organic cause for bloating and distension (such as celiac disease or other absorption disorders, intestinal dysmotility, and chronic intestinal pseudo-obstruction)
* Having alarm symptoms (weight loss, rectal bleeding, or anemia)
* Having a Body Mass Index (BMI) ≥40
* Having a history of gastrointestinal (GI) or abdominolumbopelvic surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Gastroenetrology Clinic at Ege University Hospital.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Superficial Electromyography (EMG) | At the time of the initial physiotherapist examination
  A NeuroTrac MyoPlus 4 PRO (Verity Medical LTD., UK) type EMG device will be used in the study. Bioelectrical activities of the muscles (pelvic floor muscles, abdominal muscles, diaphragm, multifidus, erector spina) will be recorded with disposable 3.2 x 3.2 cm superficial electrodes. To reduce skin impedance, the skin area will be cleaned with an alcohol swab. Active electrodes will be placed on the right side of the body, parallel to the muscle fibers, according to the reference points. The reference electrode will be placed on the anterior superior iliac spine. Measurements will be performed during six seconds of maximal voluntary contraction ('work' phase EMG activity) and sixseconds of relaxation ('rest' phase EMG activity) of the pelvic floor muscles. Measurements will be repeated for three times. The graphic and numerical data provided by the device will be recorded in the evaluation form.
Ultrasonography (USG) | At the time of the initial physiotherapist examination
  Pelvic floor displacement, bladder wall thickness and, abdominal muscles, multifidus, erector spina, diaphragma, intercostal muscle thicknesses, anorectal angle, anopubıc angle will be measured. A transabdominal diagnostic USG device (Sonospace SSI-600) with a low frequency (2-5 MHz) curvilinear transducer will be used. Muscle thickness and distance measurements will be made during frozen imaging. Muscle thickness will be measured between the upper border of the muscle fascia, which appears as a white line, and the end point of the lower border. Measurements will be taken at the expiration and during a five-second pelvic floor muscle contraction. Both measurement results will be recorded in millimeters. All measurements will be repeated three times and the average values will be noted on the evaluation form
MIP-MEP Measurement | At the time of the initial physiotherapist examination
  One of the most commonly used non-invasive methods for evaluating respiratory muscles is the measurement of Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP). These are pressures measured within the oral cavity during maximal respiration against a closed airway. MIP (Maximum Inspiratory Pressure) is the highest pressure generated to open closed alveoli at the level of residual volume (actually negative pressure). For the test, the subject is asked to perform maximum expiration, and at the end of this, the airway is occluded with a valve, prompting the individual to perform maximum inspiration and sustain it for 1-3 seconds. MEP (Maximum Expiratory Pressure), on the other hand, is the highest pressure required to deflate over-distended alveoli at the level of total lung capacity. After instructing the individual to perform maximum inspiration for MEP measurement, they are asked to perform maximum expiration against a closed airway for 1-3 seconds.
Gastrointestinal Symptom Rating Scale | At the time of the initial physiotherapist examination
  The scale evaluates how individuals have felt regarding gastrointestinal issues in the past week. The scale consists of 15 questions with 5 subscales: reflux, indigestion, diarrhea, constipation, and abdominal pain. Higher scores obtained from the scale indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No